CLINICAL TRIAL: NCT03042923
Title: Intestinal Permeability and Endometriosis
Status: Completed | Type: Observational
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Other Study IDs: 16-029
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Endometriosis
Keywords: Intestinal permeability
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment: Twenty patients, known to us through care at Women's Surgery Center and the private practice of Dr. R. Scott Furr, will be invited to enroll based on a history of pelvic pain and a plan for surgical evaluation and intervention
  Interventions: Drug: lactulose:mannitol (L:M) oral challenge
- Control: Ten healthy female patients, without pelvic pain or history of autoimmune disease, will be asked to participate as controls.
  Interventions: Drug: lactulose:mannitol (L:M) oral challenge

INTERVENTIONS:
Drug: lactulose:mannitol (L:M) oral challenge

SUMMARY:
The objective of this project will be to determine whether patients with a surgical diagnosis of endometriosis have impaired intestinal permeability as compared with healthy controls. This would suggest the presence of an environmentally triggered and intestinally mediated association in the etiology of endometriosis. This would be a proof of concept trial to establish whether there is in fact a relationship worthy of future research.

DETAILED DESCRIPTION:
Twenty patients with a clinical diagnosis of endometriosis who are scheduled for surgical evaluation will be eligible for the study arm of the research. Ten women without history of autoimmune disease or pelvic pain will serve as controls.

Study subjects will undergo testing for intestinal permeability a week or more before their scheduled surgery. Both controls and pain patients will be tested for permeability using a lactulose:mannitol (L:M) oral challenge. Each subject will ingest an oral preparation of Lactulose 5 gm, Mannitol 1gm and water. This preparation is available as a test kit through Genova Diagnostics labs. Erlanger Hospital lab does not have a test for measuring urinary excretion of L:M, or other method of assessing intestinal permeability.

Urine is collected over six hours and is then measured for ratio of L:M. An L:M ratio >0.10 is consistent with increased intestinal permeability. Normally the gut does not absorb lactulose unless permeability is present. NSAIDS and alcohol increase intestinal permeability; therefore subjects will be asked to avoid the use of NSAIDS and alcoholic beverages for a week prior to the test.

Following the L:M testing, the patients who have been enrolled will undergo surgery as planned. The surgeons should be blinded to the results of the L:M testing until after the surgery. It is assumed that some of the patients will have surgical evidence of endometriosis and some will not. The ultimate categories for analysis will be 1) Pain with biopsy proven endometriosis, and surgical staging of disease, 2) Pain without surgical evidence of endometriosis, 3) Control patients with no history of chronic pain, alcoholism, celiac disease or other autoimmune disease. As a secondary element of this study, correlation to the presence of interstitial cystitis (IC) will also be assessed as all patients in our practice who undergo surgical evaluation for chronic pain simultaneously are evaluated for IC by cystoscopy with hydrodistention.

Data that the investigators will gather includes: demographic, pelvic pain parameters, information on use of tobacco and alcohol, medical history to exclude autoimmune disease patients and patients with diabetes, intestinal permeability test results and date of test, surgical findings, American Society of Reproductive Medicine, ASRM, Endometriosis staging when applicable, presence of extrapelvic endometriosis, pathology results and presence or absence of interstitial cystitis.

Because this is an unexplored area of research, preliminary data to demonstrate potential efficacy before embarking on a prospective trial is essential.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with documented history of pelvic pain for the study arm.
* Healthy female controls without history consistent with autoimmune disease or pelvic pain

Exclusion Criteria:

* Co-morbid autoimmune disease such as Celiac disease, lupus, ankylosing spondylitis, alcoholism and diabetes which have been shown to exhibit elevated levels of Zonulin and therefore impaired intestinal permeability. Drinking alcohol and taking NSAIDS elevate intestinal permeability and would affect data.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants will be recruited through care at Women's Surgery Center and the private practice of Dr. R. Scott Furr and through Erlanger Women's Specialty Services and the practice of Dr. Shanti Mohling. Participants will be invited to enroll based on a history of pelvic pain and a plan for surgical evaluation and intervention. Ten healthy female women, without pelvic pain or history of autoimmune disease, will be asked to participate as controls.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-04; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
lactulose:mannitol (L:M) oral challenge | 6 hrs
  Urine is collected over six hours and is then measured for ratio of L:M. An L:M ratio >0.10 is consistent with increased intestinal permeability. Normally the gut does not absorb lactulose unless permeability is present.

SECONDARY OUTCOMES:
Surgical Findings | 24 hrs
  Pathology reported-- endometriosis or no endometriosis

CONTACTS AND LOCATIONS:
Overall Officials: Shanti Mohling, MD, Principal Investigator — UT College of Medicine; Patti Bush, EdD, Study Director — UT College of Medicine; Garrett Lam, MD, Study Chair — UT College of Medicine; Steve Radtke, MD, Principal Investigator — UT College of Medicine
Locations (2):
- United States (2):
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Women's Surgery Center, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WITEBSKY E, ROSE NR, TERPLAN K, PAINE JR, EGAN RW. Chronic thyroiditis and autoimmunization. J Am Med Assoc. 1957 Jul 27;164(13):1439-47. doi: 10.1001/jama.1957.02980130015004. No abstract available. PMID 13448890
- [Background] Eisenberg VH, Zolti M, Soriano D. Is there an association between autoimmunity and endometriosis? Autoimmun Rev. 2012 Sep;11(11):806-14. doi: 10.1016/j.autrev.2012.01.005. Epub 2012 Feb 4. PMID 22330229
- [Background] Fasano A. Physiological, pathological, and therapeutic implications of zonulin-mediated intestinal barrier modulation: living life on the edge of the wall. Am J Pathol. 2008 Nov;173(5):1243-52. doi: 10.2353/ajpath.2008.080192. Epub 2008 Oct 2. PMID 18832585
- [Background] Fasano A. Zonulin, regulation of tight junctions, and autoimmune diseases. Ann N Y Acad Sci. 2012 Jul;1258(1):25-33. doi: 10.1111/j.1749-6632.2012.06538.x. PMID 22731712
- [Background] Watts T, Berti I, Sapone A, Gerarduzzi T, Not T, Zielke R, Fasano A. Role of the intestinal tight junction modulator zonulin in the pathogenesis of type I diabetes in BB diabetic-prone rats. Proc Natl Acad Sci U S A. 2005 Feb 22;102(8):2916-21. doi: 10.1073/pnas.0500178102. Epub 2005 Feb 14. PMID 15710870
- [Background] Bjarnason I, MacPherson A, Hollander D. Intestinal permeability: an overview. Gastroenterology. 1995 May;108(5):1566-81. doi: 10.1016/0016-5085(95)90708-4. PMID 7729650